CLINICAL TRIAL: NCT04245839
Title: A Phase 2, Open-label, Single Arm, Multicohort, Multicenter Trial to Evaluate the Efficacy and Safety of JCAR017 in Adult Subjects With Relapsed or Refractory Indolent B-cell Non-Hodgkin Lymphoma (NHL)
Brief Title: A Study to Evaluate the Efficacy and Safety of JCAR017 in Adult Subjects With Relapsed or Refractory Indolent B-cell Non-Hodgkin Lymphoma (NHL)
Acronym: TRANSCEND FL
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JCAR017-FOL-001; U1111-1244-9768 (Other: WHO); 2024-510966-18 (Other: EU CTR)
Record Dates: First submitted 2020-01-27; First posted 2020-01-29 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Lymphoma, Non-Hodgkin
Keywords: B-cell Non-Hodgkin Lymphoma (NHL); JCAR017; Relapsed or Refractory; Follicular Lymphoma; Marginal Zone Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, B-Cell; Recurrence; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Administration of JCAR017 (Experimental): * Subjects will be treated with fludarabine IV (30 mg/m2/day for 3 days) and cyclophosphamide IV (300 mg/m2/day for 3 days) prior to JCAR017 infusion. Refer to the most recent package inserts for further details on administration of these agents.
  * JCAR017 will be infused on Day 1 at a target dose of 100 × 10^6 CAR-positive viable T cells (CAR+ T cells), 2 to 7 days after completion of LD chemotherapy. Each JCAR017 dose includes CD4+ CAR+ T cells and CD8+ CAR+ T cells.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Drug: JCAR017

INTERVENTIONS:
Drug: Fludarabine — Fludarabine
Drug: Cyclophosphamide — Cyclophosphamide
Drug: JCAR017 — JCAR017

SUMMARY:
This is a global Phase 2, open-label, single-arm, multicohort, multicenter study to evaluate efficacy and safety of JCAR017 in adult subjects with r/r FL or MZL.

The study will be conducted in compliance with the International Council on Harmonisation (ICH) of Technical Requirements for Registration of Pharmaceuticals for Human Use/Good Clinical Practice (GCP) and applicable regulatory requirements.

This study is divided into three periods:

* Pretreatment, which consists of screening assessments, leukapheresis and the Pretreatment evaluation;
* Treatment, which starts with the administration of lymphodepleting (LD) chemotherapy and continues through JCAR017 administration at Day 1 with follow-up through Day 29;
* Posttreatment, which includes follow-up assessments for disease status and safety for 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Relapsed or refractory follicular lymphoma (FL) (Grade 1, 2 or 3a) or marginal zone lymphoma (MZL) histologically confirmed within 6 months of screening, as assessed by local pathology
2. Patients should have received at least one prior therapy that includes anti-CD20 and alkylating agent
3. Follicular lymphoma patients: Received at least one prior line of systemic therapy. Patients that received one prior line of systemic therapy are eligible if they present with high risk features. Patients that received two or more prior lines of systemic therapy are eligible, assuming one of the prior lines includes anti-CD20 and alkylating agent (as listed in criterion 2)
4. Marginal zone lymphoma patients: Received two or more prior lines of systemic therapy, assuming one of the prior lines includes anti-CD20 and alkylating agent (as listed in criterion 2) or relapsed after hematopoietic stem cell transplant
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
6. Adequate organ function
7. Adequate vascular access for leukapheresis procedure

Exclusion Criteria:

1. Evidence or history of composite Diffuse large B-cell lymphoma (DLBCL) and FL, or of transformed FL
2. WHO subclassification of duodenal-type FL
3. Central nervous system-only involvement by malignancy (subjects with secondary central nervous system (CNS) involvement are allowed on study)
4. History of another primary malignancy that has not been in remission for at least 2 years, with the exception of non-invasive malignancies
5. Prior CAR T-cell or other genetically-modified cell therapy
6. History of or active human immunodeficiency virus (HIV)
7. Active hepatitis B or active hepatitis C
8. Uncontrolled systemic fungal, bacterial, viral or other infection despite appropriate antibiotics or other treatment
9. Active autoimmune disease requiring immunosuppressive therapy
10. Presence of acute or chronic graft-versus-host=disease
11. History of significant cardiovascular disease
12. History or presence of clinically relevant central nervous system pathology
13. Allogenic-hematopoietic stem cell transplant (Allo-HSCT) within 90 days of leukapheresis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Estimated)
Dates: Start 2020-07-14 (Actual); Primary Completion 2031-09-30 (Estimated); Study Completion 2031-09-30 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Up to 60 months
  Is defined as the percentage of participants achieving either a partial response (PR) or complete response (CR) at any time up to 60 months after JCAR017 treatment as assessed by PET-CT and/or CT using "The Lugano classification"

SECONDARY OUTCOMES:
Complete response rate (CRR) as assessed but PET-CT and/or CT using "The Lugano Classification" | Up to 60 months
  Is defined as the percentage of subjects achieving a CR at any time up to 60 months after JCAR017 treatment
Duration of Response (DOR) if Best Overall Response (BOR) is CR, as assessed by PET-CT and/or CT using "The Lugano Classification" | Up to 60 months
  is defined for subjects with a BOR of CR as the time from first response (CR or PR) to disease progression or death from any cause up to 60 months after JCAR017 treatment
Duration of Response (DOR) as assessed by PET-CT and/or CT using "The Lugano Classification" | Up to 60 months
  is defined as the time from first response (CR or PR) to disease progression or death from any cause, whichever occurs first up to 60 months after JCAR017 treatment
Progression-Free Survival (PFS) as assessed by PET-CT and/or CT using "The Lugano Classification" | Up to 60 months
  is defined as the time from start of JCAR017 to disease progression or death from any cause, whichever occurs first up to 60 months after JCAR017 treatment
Overall Survival (OS) | Up to 60 months
  is defined as the time from start of JCAR017 to time of death due to any cause up to 60 months after JCAR017 treatment
Adverse Events (AEs) | Up to 60 months
  An AE is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a subject during the course of a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the subject's health, including laboratory test values, regardless of etiology. Any worsening (ie, any clinically significant adverse change in the frequency or intensity of a preexisting condition) should be considered an AE.
Pharmacokinetics - Cmax | Up to 60 months
  Maximum concentration
Pharmacokinetics - Tmax | Up to 60 months
  Time to maximum concentration
Pharmacokinetics - AUC | Up to 60 months
  Area under the curve
European Organization for Research and Treatment of Cancer - Quality of Life C30 questionnaire (EORTC QLQ-C30) | Up to 24 months
  is questionnaire that will be used as a measure of health-related quality of life.
  The EORTC QLQ-C30 is composed of both multi-item scales and single item measures. These include five functional scales (physical, role, emotional, cognitive and social), three symptom scales (fatigue, nausea/vomiting, and pain), a global health status/health-related quality of life (HRQoL) scale, and six single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). Each of the multi-item scales includes a different set of items - no item occurs in more than one scale.
Functionality Assessment of Cancer Therapy Lymphoma Subscale (FACT-LymS) | Up to 24 months
  is a 15-item lymphoma-specific additional concerns subscale. This subscale addresses symptoms and functional limitations are important to lymphoma patients. The FACT-LymS items are scored on a 0 ("Not at all") to 4 ("Very much") response scale. Items are aggregated to a single score on a 0-60 scale. High scores indicate lower symptom burden.

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (49):
- United States (23):
  - Local Institution - 111, Santa Monica, California
  - Local Institution - 107, Aurora, Colorado
  - Local Institution - 105, New Haven, Connecticut
  - Local Institution - 103, Chicago, Illinois
  - Local Institution - 109, Niles, Illinois
  - Local Institution - 122, Iowa City, Iowa
  - Local Institution - 124, Wichita, Kansas
  - Local Institution - 102, Baltimore, Maryland
  - Local Institution - 100, Boston, Massachusetts
  - Local Institution - 101, Boston, Massachusetts
  - Local Institution - 127, Detroit, Michigan
  - Local Institution - 123, Morristown, New Jersey
  - Local Institution - 116, New York, New York
  - Local Institution - 110, Charlotte, North Carolina
  - Local Institution - 112, Cleveland, Ohio
  - Local Institution - 114, Portland, Oregon
  - Local Institution - 117, Philadelphia, Pennsylvania
  - Local Institution - 113, Sioux Falls, South Dakota
  - Local Institution - 121, Dallas, Texas
  - Local Institution - 104, Houston, Texas
  - Local Institution - 119, Houston, Texas
  - Local Institution - 115, Charlottesville, Virginia
  - Local Institution - 108, Seattle, Washington
- Local Institution - 450, Vienna, Austria
- Canada (2):
  - Local Institution - 150, Toronto, Ontario
  - Local Institution - 151, Montreal, Quebec
- France (6):
  - Local Institution - 252, Lille
  - Local Institution - 251, Montpellier
  - Local Institution - 255, Paris
  - Local Institution - 250, Pierre-Bénite
  - Local Institution - 253, Rennes
  - Local Institution - 254, Toulouse
- Germany (5):
  - Local Institution - 500, Ulm, Baden-Wurttemberg
  - Local Institution - 504, Regensburg, Bavaria
  - Local Institution - 501, Cologne
  - Local Institution - 503, Karlsruhe
  - Local Institution - 502, Munich
- Italy (2):
  - Local Institution - 300, Bergamo
  - Local Institution - 301, Naples
- Japan (4):
  - Local Institution - 553, Sapporo, Hokkaido
  - Local Institution - 550, Chuo-ku, Tokyo
  - Local Institution - 551, Minato-ku, Tokyo
  - Local Institution - 552, Fukuoka
- Spain (3):
  - Local Institution - 353, Madrid
  - Local Institution - 350, Salamanca
  - Local Institution - 351, Seville
- Local Institution - 600, Stockholm, Sweden
- United Kingdom (2):
  - Local Institution - 200, London
  - Local Institution - 201, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Information relating to our policy on data sharing and the process for requesting data can be found at the following link:
  https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- [Derived] Morschhauser F, Dahiya S, Palomba ML, Martin Garcia-Sancho A, Reguera Ortega JL, Kuruvilla J, Jager U, Cartron G, Izutsu K, Dreyling M, Kahl B, Ghesquieres H, Ardeshna K, Goto H, Barbui AM, Abramson JS, Borchmann P, Fleury I, Mielke S, Skarbnik A, de Vos S, Kamdar M, Karmali R, Viardot A, Farazi T, Fasan O, Lymp J, Vedal M, Nishii R, Avilion A, Papuga J, Kumar J, Nastoupil LJ. Lisocabtagene maraleucel in follicular lymphoma: the phase 2 TRANSCEND FL study. Nat Med. 2024 Aug;30(8):2199-2207. doi: 10.1038/s41591-024-02986-9. Epub 2024 Jun 3. PMID 38830991
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT04245839.html